CLINICAL TRIAL: NCT01809925
Title: Randomized, Double-blind, Placebo-controlled, 2-treatment, 3-period Crossover Design Study of the Efficacy and Tolerability of Psyllium 6.8 g Provided as Sugarfree Metamucil® Fiber Supplement Powder Versus Placebo on Satiety in Healthy Volunteers
Brief Title: Study of Psyllium 6.8 g Versus Placebo on Satiety in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012126
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2013-03

CONDITIONS: Hunger
MeSH Terms: interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- psyllium fiber 6.8g (Experimental): Two (2) packets Metamucil Orange Sugar Free Fiber Singles (psyllium 6.8 g) thoroughly mixed in Ten (10) ounces of water. Subjects will drink their assigned test product as quickly as possible immediately before eating breakfast at each visit.
  Interventions: Dietary Supplement: psyllium fiber 6.8g
- placebo (Placebo Comparator): One (1) level teaspoon of placebo product thoroughly mixed in Ten (10) ounces of water. Subjects will drink their assigned test product as quickly as possible immediately before eating breakfast at each visit.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: psyllium fiber 6.8g — Subjects will drink their assigned test product as quickly as possible immediately before eating breakfast at each visit.
  Other Names: Metamucil Orange Sugar Free Fiber Singles (psyllium 6.8 g)
  Arms: psyllium fiber 6.8g
Dietary Supplement: placebo — Subjects will drink their assigned test product as quickly as possible immediately before eating breakfast at each visit.
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-treatment, 3-period crossover design study to evaluate the effects of psyllium 6.8 g provided as sugarfree Metamucil fiber supplement powder dissolved in water versus placebo on satiety measures in healthy volunteers. This study will be conducted at a single study site.

DETAILED DESCRIPTION:
A total of 45 subjects will be enrolled in this study. Approximately equal numbers of men and women will be enrolled, with a race distribution consistent with the US population. Eligible subjects will be randomly assigned to 1 of 2 test product sequences at Test Period 1 (Visit 2) using a block randomization. Subjects will participate in 3 test periods (Test Period 1, Visits 2-4; Test Period 2, Visits 5-7; and Test Period 3, Visits 8-10) and will receive test product once a day before breakfast for 3 days within each period. Test periods will be separated by a minimum 4-day washout period in which no test product will be administered.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible to participate in the study:

* routinely eat breakfast daily;
* agree to eat 100% of the food provided during the study, drink 10 ounces of water with the test product immediately before breakfast, and only eat a light snack after dinner before fasting overnight beginning at 10:00 PM prior to the next visit;
* have a screening VAS Hunger score > 50 before eating breakfast that moves towards less hunger after eating breakfast;
* have 1-2 bowel movements per day that are typically rated as 3, 4, or 5 on the Bristol Stool Form Scale;
* in good general health based on medical history;
* if female, be postmenopausal or if of child-bearing capacity agree to use an adequate form of contraception (eg, surgical sterilization, birth control pills, birth control implants, condoms AND spermicide, abstinence);
* have a body mass index (BMI) ≥ 18.5 but < 28 kg/m2;
* able to fulfill the requirements of the protocol and provide written consent;
* willing to abstain from any weight control or satiety supplements during the study;
* willing to refrain from taking any psyllium containing products or fiber supplements during the study with the exception of the test products;
* willing to maintain lifestyle habits for the duration of the study (eg, do not change exercise habits or begin a weight loss diet);
* willing to refrain from exercise on the mornings prior to arriving at the study site;
* willing to abstain from alcohol for 2 days prior to the first day of each test period through the last day of each test period;
* willing not to consume caffeine for 24 hours prior to the first day of each test period through the last day of each test period.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* have any history of heart, liver, kidney, nerve, blood disorder, or cancer(except for treated basal cell cancer with a documented 6-month remission), or metabolic, hormone, or gastrointestinal (GI) disease;
* have a history of an eating disorder;
* have difficulty swallowing;
* have a history of gastrointestinal surgery (except appendectomy) or gastrointestinal bleeding;
* are currently alcohol or chemically dependent (a urine test for drugs of abuse will be given);
* report use of tobacco, smoking cessation products, or products containing nicotine within 3 months;
* have a significant psychiatric disorder;
* any use of prescription drugs, with the exception of birth control pills, within 14 days prior to the study or antibiotics in the past 30 days;
* any use of non-prescription drugs within 7 days prior to the study;
* used psyllium containing products or fiber supplements within the past month;
* have a history of phenylketonuria (PKU);
* have a history of a severe allergic reaction to psyllium;
* are currently on a structured formal diet (eg, Jenny Craig, Atkins);
* typically drink more than 70 ounces of liquid during the day (ie, approximately 4 bottles of water, each 16.9 ounces)
* have a history or presence, upon clinical evaluation, of any illness or condition that might impact the safety of the study product;
* participated in a clinical drug study or used an investigational new drug within 30 days of dosing;
* pregnant or nursing, if female;
* engage in excessive exercise that is extreme in frequency or duration;
* find the study meals unpalatable

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
satiety (VAS Hunger 3-day average) | Hours 0-4.5
  VAS Hunger 3-day average. This endpoint will be calculated by averaging all evaluable post-breakfast scores across Days 1, 2, and 3. VAS Hunger is assessed on a horizontal 100-mm VAS anchored on the left by the phrase "Not at all hungry" (score = 0) and on the right by "As hungry as I have ever felt" (score = 100).

SECONDARY OUTCOMES:
Satiety Labeled Intensity Magnitude (SLIM) 3-day average | Hours 0-4.5
  SLIM 3-day average is calculated by averaging all evaluable post-breakfast scores across Days 1, 2, and 3. SLIM scale gauges perceived hunger/fullness following a meal using 11 phrases placed along a vertical line scale anchored at the bottom by "Greatest imaginable hunger" (score = -100) and at the top by "Greatest imaginable fullness" (score = 100).
VAS Desire to Eat 3-day average | Hours 0-4.5
  The VAS Desire to Eat 3-day average is calculated by averaging all evaluable post-breakfast scores across Days 1, 2, and 3. The VAS Desire to Eat Scale asks subjects to rate their desire to eat using a horizontal 100-mm VAS anchored on the left by the phrase "No desire at all" (score = 0) and on the right by "As strong as I have ever felt" (score = 100)
VAS Hunger 3-day average for hours 3.0 - 4.5 | Hours 3.0 - 4.5
  The VAS Hunger 3-day average for hours 3.0 - 4.5 is calculated by averaging all evaluable post-breakfast scores for hours 3.0, 3.5, 4.0, and 4.5 across Days 1, 2, and 3. The VAS Desire to Eat Scale asks subjects to rate their desire to eat using a horizontal 100-mm VAS anchored on the left by the phrase "No desire at all" (score = 0) and on the right by "As strong as I have ever felt" (score = 100).
SLIM 3-day average for Hours 3.0-4.5 | Hours 3.0-4.5
  SLIM 3-day average for Hours 3.0-4.5 is calculated by averaging all evaluable post-breakfast scores for hours 3.0, 3.5, 4.0, and 4.5 across Days 1, 2, and 3. The SLIM scale gauges perceived hunger/fullness following a meal using 11 phrases placed along a vertical line scale anchored at the bottom by "Greatest imaginable hunger" (score = -100) and at the top by "Greatest imaginable fullness" (score = 100).
VAS Desire to Eat 3-day average for hours 3.0 - 4.5 | Hours 3.0-4.5
  The VAS Desire to Eat 3-day average for hours 3.0-4.5 is calculated by averaging all evaluable post-breakfast scores for hours 3.0, 3.5, 4.0, and 4.5 across Days 1, 2, and 3. The VAS Desire to Eat Scale asks subjects to rate their desire to eat using a horizontal 100-mm VAS anchored on the left by the phrase "No desire at all" (score = 0) and on the right by "As strong as I have ever felt" (score = 100).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Brum, MD, Study Director — Procter and Gamble
Locations (1):
- Study Center, Cincinnati, Ohio, United States